CLINICAL TRIAL: NCT07044843
Title: Oxygen Therapy During Exercise Training in Inpatient Rehabilitation in Chronic Lung Disease- Does it Matter?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: inRehaExO2_normoxia_hyperoxia
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: COPD
Keywords: Oxygen; Exercise; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia (Sham Comparator): Sham air (ambient air) (5l/min) will be applied with the oxygen concentrator EverFloTM via nasal cannula.
  Interventions: Other: Standard ambiant air will be breathed during endurance training.
- Hyperoxia (Active Comparator): Standardized supplemental oxygen therapy (SSOT) (5l/min) will be applied with the oxygen concentrator EverFloTM via nasal cannula during training
  Interventions: Other: Oxygen
- Hypoxia (Experimental): This group will train at moderate altitude.
  Interventions: Other: Standard ambiant air will be breathed during endurance training.

INTERVENTIONS:
Other: Oxygen — SSOT and sham air (5l/min) will be applied with the oxygen concentrator EverFloTM via nasal cannula during training
  Arms: Hyperoxia
Other: Standard ambiant air will be breathed during endurance training. — ambiant air
  Arms: Hypoxia; Normoxia

SUMMARY:
The aim of the current study is the effect of SSOT during a 3-weeks inpatient pulmonary rehabilitation program. Further aim is to analyze exercise endurance, distinguishing between those exercising whilst breathing air at 760m "normoxia", breathing air at approx. 1600m "hypoxia", or breathing SSOT at 760m "hyperoxia" conditions during inpatient pulmonary rehabilitation.

The objective of the study is to provide long-awaited data concerning the use of SSOT during training. To date, it is not clear whether patients with chronic lung diseases who reveal a SpO2 > 88% at rest but desaturate during exercise and thus may not qualify for long-term oxygen therapy undergoing PR benefit from supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* stable condition > 3 weeks (e.g. no exacerbations)
* resting SpO2 ≥ 88% and exercise induced hypoxemia defined by a fall in SpO2 by ≥ 4% and/or below 90% during a 6-minute walk test (6MWT)
* informed consent as documented by signature.

Exclusion Criteria:

* Severe daytime resting hypoxemia (SpO2 < 88%)
* long-term oxygen therapy
* unstable condition requiring adaptation of pharmacologic and other treatment modalities or requirement of intensive care or relevant severe concomitant disease
* inability to follow the procedures of the study, e.g. due to language problems psychological disorders, neurological or orthopedic problems with walking disability or inability to ride a bicycle
* women who are pregnant or breast feeding
* enrolment in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cycling CWRET time normoxia vs hypoxia vs hyperoxia | from baseline to 3 weeks

SECONDARY OUTCOMES:
6 minute walk test (6MWT) | 3 weeks
  6 minute walk distance (6MWD), SpO2 and heart rate at the end of the 6 minute walk test (6MWT) from baseline to 3 weeks at normoxia vs hypoxia vs hyperoxia
Hospital Anxiety and Depression Scale (HADS) normoxia vs hypoxia vs hyperoxia | 3 weeks
  HADS-A (Anxiety): 7 items
  HADS-D (Depression): 7 items
  Each item is scored from 0 to 3, resulting in:
  Minimum score per subscale: 0
  Maximum score per subscale: 21
  Interpretation:
  Higher scores indicate worse psychological status.
  Scores of 0-7: Normal
  Scores of 8-10: Borderline abnormal
  Scores of 11-21: Abnormal (clinically relevant anxiety or depression)
mMRC score at normoxia vs hypoxia vs hyperoxia | 3 weeks
  The scale ranges from 0 to 4.
  Each grade reflects a different level of functional limitation due to dyspnea.
  Minimum score: 0 Maximum score: 4
  Interpretation:
  Higher scores indicate more severe dyspnea (worse outcome).
CAT score (COPD assessments tool) normoxia vs hypoxia vs hyperoxia | 3 weeks
  It consists of 8 items, each scored from 0 to 5.
  The total score ranges from:
  Minimum score: 0 Maximum score: 40
  Interpretation:
  Higher scores indicate greater symptom burden and worse health status.
  Score bands for interpretation:
  0-10: Low impact
  11-20: Medium impact
  21-30: High impact
  31-40: Very high impact
Chronic respiratory questionnaire (CRQ) normoxia vs hypoxia vs hyperoxia | 3 weeks
  The CRQ consists of 20 items across four domains:
  Dyspnea (5 items)
  Fatigue (4 items)
  Emotional function (7 items)
  Mastery (4 items)
  Each item is scored on a 7-point Likert scale:
  Minimum score per item: 1
  Maximum score per item: 7
  Interpretation:
  Higher scores indicate better health-related quality of life (less impairment).
  Mean scores are calculated per domain and as a total score.
Change in cycling CWRET time normoxia vs hypoxia vs hyperoxia | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- National center for cardiology and internal medicine, Bishkek, Kyrgyzstan
- Eastern Switzerland University of Applied Sciences, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
individual patient data will be shared upon personal request to the corresponding author